CLINICAL TRIAL: NCT05738720
Title: The Effect of Close Follow-Up Home Based Pulmonary Rehabilitation on Exacerbation Frequency and Hospital Admission in Severe COPD Cases
Brief Title: Effect of Home Based Pulmonary Rehabilitation on Exacerbation and Hospital Admission in Severe COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, ESRA PEHLIVAN, Assoc. Prof. Dr., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Homespirometry1
Record Dates: First submitted 2023-01-15; First posted 2023-02-22 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: COPD Exacerbation
Keywords: copd exacerbation; pulmonary rehabilitation; spirometry; hospital admission

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Homespirometer Group (HsGr) (Experimental): Patients will be taught to use the homespirometer device, download the phone application, use the application, use the video call feature, measure saturation and heart rate with the same device, and daily symptom scoring in the device's system.
  Patients will be asked to perform pulmonary function tests with a spirometer device, measure saturation and heart rate, score symptoms, and write down any problems related to their illness twice a week on days without exercise. The evaluations made after 2 tests. They will be sent to the researchers via the device.andthe video containing the exercises after the first training will be sent to them via whatsapp for the exercise compliance of the patients. In the first exercise week, the first 2 exercise sessions will be done one-on-one via video call, and the exercises will be done correctly.
  Interventions: Device: Teknikel Spirobank Home Type Respiratory Function Tester (Homespirometer); Other: Exercise Programme
- Control Group (CGr) (Active Comparator): The same exercise training will be taught to the study group and the same exercise video will be sent to the patients via WhatsApp. The first 2 exercise sessions will be done one-on-one via video call (via whatsapp), and the exercises will be done correctly. Patients will be given an exercise diary and asked to take notes on their weekly exercises.
  Interventions: Other: Exercise Programme

INTERVENTIONS:
Device: Teknikel Spirobank Home Type Respiratory Function Tester (Homespirometer) — Pulmonary Function Test (PFT): Pulmonary function test will be performed with a Teknikel Spirobank home pulmonary function test device. In the study group, the patient will make weekly measurements at home and send it to the physiotherapist. In the control group, evaluation will be made with the device only at the beginning and end of the treatment.
  Arms: Homespirometer Group (HsGr)
Other: Exercise Programme — Exercise Program
  * Breathing exercises: Chest, diaphragmatic breathing and lower basal breathing exercises will be performed with 10 repetitions.
  * Resistance exercises: Strengthening exercises will be performed on the major muscle groups of the upper and lower extremities by using medium hardness therabant. During the exercises, the patient's fatigue and dyspnea levels will be questioned using the Borg scale, and breaks will be given when necessary. The exercises will be performed with a medium-hardness therabband. Exercises will be given for the upper extremity and lower extremity, and the patients will be asked to do 10 repetitions.
  * Gait training: In line with the data obtained from the 6-minute walking test, gait training will be given on flat ground at 60% workload (land-based walking). Patients will be allowed to walk on flat ground at 60% workload, at a time calculated based on the results of the 6-minute walk test.

SUMMARY:
The study is a randomized controlled trial. The cases will be divided into two groups as the Homespirometer group and the control group. Breathing exercises, aerobic exercise and peripheral muscle strengthening will be performed in both groups. A home-type spirometer will be given to the homespirometer group and it will be requested to send the spirometric measurement every week. The cases will be called to the hospital for control and evaluated at baseline, 3rd, 6th and 12th months. Evaluations include assessments such as exercise capacity measurement, muscle strength measurement, disease attack frequency, symptom scoring.

DETAILED DESCRIPTION:
Pulmonary Rehabilitation (PR) is a comprehensive intervention designed to improve not only exercise, education and behavioral changes, but also the physical and psychological state of individuals, based on detailed patient evaluation and subsequent patient-specific therapies in individuals with chronic respiratory disease. It is integrated into the lifelong care and management of the chronic respiratory patient. It requires an active collaboration between the patient, family, and the Pulmonary Rehabilitation team. Due to the complex nature of respiratory diseases, many disciplines should be involved in the maintenance of treatment.

Pulmonary rehabilitation is a useful treatment component in almost all chronic respiratory patients, especially COPD (Chronic obstructive pulmonary disease). There are studies showing that it reduces the number of attacks and the frequency of hospitalization even in COPD patients with frequent attacks. As pulmonary rehabilitation methods; It is possible to see that there are many types such as supervised exercise programs in the hospital, telephone monitoring or home programs.In-hospital supervised programs are time-consuming and costly applications. This situation causes an increase in the tendency towards applications without direct supervision and increases the need for studies on the effectiveness and benefits of these applications.

The use of home-type spirometers are practical devices that provide close monitoring of respiratory functions and enable the detection of disease symptoms in a short time. The use of these devices has increased especially during the pandemic period. In a study conducted with asthma patients, it was reported that early diagnosis and intervention is possible in cases with self-monitoring by mobile spirometry. In another study, in which e-monitoring of cases with duchenne muscular dystrophy (DMD) was performed with a spirometer device during the covid 19 pandemic, the importance of regular spirometric follow-ups of DMD cases as a part of their daily routine and making it a part of health care services was emphasized.

In our study, advanced stage COPD cases constitute the case group. The exacerbation and hospital admission rates are extremely high in these patients. There are also transfer problems to the hospital due to existing physical limitations. With the planned study, close follow-up of the patients with the help of home-type spirometry will be carried out over a 1-year period, and a pulmonary rehabilitation exercise program will be applied in this process. The effect of the applied follow-up and exercise program on disease exacerbation and hospital admission rates will be examined.

ELIGIBILITY:
Inclusion Criteria:

Being between the ages of 18-75

* Having a diagnosis of COPD stages C and D diagnosed according to the GOLD (Global Initiative for Chronic Obstructive Lung Disease) clinical diagnostic criteria
* Presence of dyspnea on exertion
* Stable clinical condition at the time of inclusion without infection or exacerbation in the previous 4 weeks
* Having the ability to use a smart phone and spirometer after training

Exclusion Criteria:

* Patients with severe comorbid diseases, unstable coronary artery disease, collagen vascular diseases and needing high flow oxygen therapy (˃ 3-4 L \min).
* A history of effort-related syncope or any comorbidity (such as severe orthopedic or neurological deficits or unstable heart disease) that precludes exercise training.
* Participation in a pulmonary rehabilitation program within the past 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Number of exacerbations follow-up | 1 month after the evaluation
  After the first evaluation, he will be questioned at the 1st month follow-ups. Apart from this, patients will be asked to write in the notes section and contact the researchers in case of exacerbation through the spirometer device.
Number of hospital admissions | 1 month after the evaluation
  After the first evaluation, he will be questioned at the 1st month follow-ups. Apart from this, patients will be asked to write in the notes section and contact the researchers in case of exacerbation through the spirometer device.
Number of exacerbations follow-up | 3 month after the first evaluation
  After the first evaluation, he will be questioned at the 3rd month follow-ups. Apart from this, patients will be asked to write in the notes section and contact the researchers in case of exacerbation through the spirometer device.
Number of exacerbations follow-up | 6 month after the first evaluation
  After the first evaluation, he will be questioned at the 6th month follow-ups. Apart from this, patients will be asked to write in the notes section and contact the researchers in case of exacerbation through the spirometer device.
Number of exacerbations follow-up | 12 month after the first evaluation
  After the first evaluation, he will be questioned at the 12th month follow-ups. Apart from this, patients will be asked to write in the notes section and contact the researchers in case of exacerbation through the spirometer device.
Number of hospital admissions | 3 month after the first evaluation
  After the first evaluation, he will be questioned at the 3rd month follow-ups. Apart from this, patients will be asked to write in the notes section and contact the researchers in case of exacerbation through the spirometer device.
Number of hospital admissions | 6 month after the first evaluation
  After the first evaluation, he will be questioned at the 6th month follow-ups. Apart from this, patients will be asked to write in the notes section and contact the researchers in case of exacerbation through the spirometer device.
Number of hospital admissions | 12 month after the first evaluation
  After the first evaluation, he will be questioned at the 12th month follow-ups. Apart from this, patients will be asked to write in the notes section and contact the researchers in case of exacerbation through the spirometer device.

SECONDARY OUTCOMES:
Pulmonary Function Test (PFT) with home spirometry for FVC (Forced Vital Capacity) value | Baseline to one year
  Pulmonary function test will be performed with Teknikel Spirobank home type pulmonary. The FVC value will be calculated.
Daily Saturation Monitoring | Baseline to one year
  Saturation monitoring can be done in the PFT device. The patient will be asked to take measurements twice a week (on the specified days) and record them on the device.
Symptom scoring | Baseline to one year
  Questions about the symptomatic situation will be requested to be answered within the PFT device. The questions include questioning dyspnea and fatigue with a 3-point Likert scale. While 3 points define increased dyspnea or fatigue with 3 points, symptoms expected to decrease as they approach 0 points.
Peripheral muscle strength measurement | Baseline to one year
  The muscle groups to be tested are: (shoulder flexors, elbow flexors, hand grip, hip flexors, knee extensors and dorsi flexors. The test will be done by Lafayette brand digital muscle strength meter.
6 minutes walking test | Baseline to one year
  It will be carried out in the 30 meter corridor in accordance with ATS (American Thoracic Society) and ERS (European Respiratory Society) guidelines.
Modified medical Council Dyspnea score | Baseline to one year
  The scale is a score that measures the reflections of dyspnea degrees ranging from 0 to 4 on activities of daily living. While scoring, the patients were asked to mark the activity level that caused dyspnea in them. On this scale, 1 point defines the best condition in terms of dyspnea, and 5 points the worst.
Determination of quality of life | Baseline to one year
  The Saint George Respiratory Questionnaire (SGRQ) will be used. All of the patients will be answered the questions themselves and scores will be calculated using the score calculation algorithm (SGRQ manual version 2). The total score ranges from 0-100. A score of zero indicates normal and a score of 100 indicates maximum disability.
Psychological status assessment | Baseline to one year
  The Hospital Anxiety and Depression Scale will be used. By adding the subscale scores of the questionnaire, 0-21 points can be obtained from each of the Depression and Anxiety subscales. It is stated that 0-7 points for each subscale are in the normal range, 8-10 points suggest the presence of a mood disorder, and a score of 11 and above indicates possible mood disorder.
Cognitive status assessment | Baseline to one year
  The Montreal Cognitive Assessment (MOCA) questionnaire will be used. The highest score that can be obtained from the test is 30. A score of 21 and above is considered "normal".
Physical activity level | Baseline to one year
  The short form of the International Physical Activity Questionnaire-Short Form (IPAQ-SF) will be used. ollowing the IPAQ guidelines, the respondents will be categorized as engaged in vigorous physical activity, moderate physical activity, or low physical activity. MET-Minute (Metabolic Equivalent of Task-Minute) is calculated by multiplying the minute of activity with the MET score. When classifying populations categorically, there are three levels of physical activity identified - 'inactive', 'minimally active' and 'very active (physical activity that increases well-being)'. The 'very active' category falls on the higher threshold of activity.
Heart Rate Monitoring | Baseline to one year
  Heart rate monitoring can be done in the PFT device. The patient will be asked to take measurements twice a week (on the specified days) and record them on the device.
Pulmonary Function Test (PFT) with home spirometry for FEV1 (Forced Expiratory Volume First Second) value | Baseline to one year
  Pulmonary function test will be performed with Teknikel Spirobank home type pulmonary. The FEV1 value will be calculated.
Pulmonary Function Test (PFT) with home spirometry for FEV1/FVC (Tiffeneau indeksi) value | Baseline to one year
  Pulmonary function test will be performed with Teknikel Spirobank home type pulmonary. The FEV1/FVC value will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Esra PEHLİVAN, Assoc. Prof., Principal Investigator — Saglik Bilimleri Universitesi; Erdoğan ÇETİNKAYA, Prof. Dr., Study Director — Saglik Bilimleri Universitesi; Mustafa ÇÖRTÜK, Assoc. Prof., Study Chair — SBU Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital; Fulya Senem KARAAHMETOĞLU, M. Sc., Study Chair — Saglik Bilimleri Universitesi; Zeynep Betül ÖZCAN, M. Sc., Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- SBU Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)